CLINICAL TRIAL: NCT02061527
Title: Immediate Breast Reconstruction With or Without the Use of Acellular Dermal Matrix: A Randomized Controlled Multicenter Study
Brief Title: Breast Reconstruction With Acellular Dermal Matrix in the Setting of Breast Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other); LifeCell (Industry)
Responsible Party: Principal Investigator, Fredrik Lohmander, Fredrik Lohmander MD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FL/KUH-ADM-LFC-2014
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: ADM; Strattice; Breast reconstruction; Immediate breast reconstruction; IBR; Acellular dermal matrix; Biological mesh; Randomized controlled trial; RCT; Breast cancer; Implants; Mastectomy; Direct-to-implant
MeSH Terms: conditions — Breast Neoplasms | interventions — Plastic Surgery Procedures; strattice; Drug Implants; Mastectomy; Tissue Expansion Devices; Mammaplasty; Mastectomy, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breast reconstruction with ADM (Experimental): Implant based Breast Reconstruction with ADM. Both arms will undergo skin or nipple sparing mastectomy and immediate breast reconstruction with implants. Patients in group B with ADM and partial submuscular coverage.
  Interventions: Procedure: Reconstruction with ADM.; Procedure: Skin or nipple sparing mastectomy; Procedure: Reconstruction with implant; Procedure: Partial submuscular coverage
- Breast reconstruction without ADM (Active Comparator): Breast reconstruction without ADM. Both arms will undergo skin or nipple sparing mastectomy and immediate breast reconstruction with implant. Patients in group B will be reconstructed with implant and total submuscular coverage.
  Interventions: Procedure: Skin or nipple sparing mastectomy; Procedure: Reconstruction with implant; Procedure: Total submuscular coverage

INTERVENTIONS:
Procedure: Reconstruction with ADM. — If the patient wishes to undergo immediate implant based reconstruction, and meets the selection criteria for entering the study, she is randomly selected to be treated according to Group A or Group B. Group A (no intervention) will be reconstructed with expander or anatomical gel implant without ADM, using complete muscle coverage. Group B (Intervention) will be reconstructed with expander or anatomical gel implant using partial muscle coverage in conjunction with ADM.
  Other Names: Strattice; ADM; Implant; Immediate breast reconstruction; Acellular dermal matrix; Mastectomy; Breast cancer; Direct-to-implant; Expander; Breast reconstruction
  Arms: Breast reconstruction with ADM
Procedure: Skin or nipple sparing mastectomy — Mastectomy for invasive or pre-invasive breast cancer
  Other Names: Mastectomy; Skin sparing mastectomy; Nipple sparing mastectomy; Acellular dermal matrix; Immediate breast reconstruction; ADM; Breast cancer; Strattice; Implant
Procedure: Reconstruction with implant — Immediate breast reconstruction with implant
  Other Names: Implant; Mastectomy; Acellular dermal matrix; Direct-to-implant; Immediate breast reconstruction; ADM; Strattice; Breast cancer
Procedure: Total submuscular coverage — Implant based breast reconstruction with total submuscular coverage
  Arms: Breast reconstruction without ADM
Procedure: Partial submuscular coverage — Implant based breast reconstruction with partial submuscular coverage
  Arms: Breast reconstruction with ADM

SUMMARY:
To evaluate breast reconstruction with implants using biological mesh (Strattice™) in the setting of breast cancer treatment.

DETAILED DESCRIPTION:
OBJECTIVES: To evaluate the outcome of immediate breast reconstruction with Acellular Dermal Matrix (Strattice™), measuring safety, effectiveness, and costs. The primary outcome measure is number of unplanned surgical procedures.

STUDY DESIGN: A prospective randomized multicenter trial. One hundred and twenty patients with breast cancer will be enrolled into the study. Study duration will be two years from time of primary cancer surgery.

TRIAL DESIGN This is a randomized controlled multicenter trial, comparing IBR without (group A) and with (group B) the use of ADM. Participants eligible for the study are patients with breast cancer, planned for mastectomy, who wishes IBR with implants. Each participant is individually randomized to either be reconstructed using implants with total submuscular coverage (A) or reconstruction with ADM and partial muscle coverage (B).

Method of assigning patients to treatment groups:

After signing and dating the informed consent the patient is entered into the study. If all inclusion and none of the exclusion criteria are full filled, the patient will be randomized to group A or group B.

TREATMENT/ INTERVENTION The decision and treatment plan advocating mastectomy is based on multi disciplinary conference (MDT), and the diagnosis of invasive or pre-invasive (in situ) breast cancer is made on triple assessment. If the patient wishes to undergo immediate implant based reconstruction, and meets the selection criteria for entering the study, she is randomly selected to be treated according to Group A or Group B. Group A will be reconstructed with expander or anatomical gel implant without ADM, using complete muscle coverage. Group B will be reconstructed with expander or anatomical gel implant using partial muscle coverage in conjunction with ADM.

Randomization at enrollment is made with regard to the use of ADM or not, so both expander and direct-to-implant techniques will be utilized in both groups, depending on the quality of skin flaps at time of surgery.

RANDOMIZATION TYPE Patients will be allocated to treatment according to permuted block technique. The actual randomization will be performed using computer based system located at Regional Cancer Center (RCC) within Karolinska Institutet. In this system inclusion and exclusion criteria will be automatically checked before patients are randomized to treatment. The randomization process will be stratified for the participating units.

STATISTICAL METHODS The main endpoint to be analyzed is the proportion of unplanned reoperations after the initial breast reconstruction. The difference in proportions between the two groups will be presented as a difference in proportion together with a 95% confidence interval. Differences will be tested using Fishers Exact Test. Logistic regression will be used to take into account possible confounding factors.

STUDY MANAGEMENT Data recording: The investigators will ensure that all data from patient visits are entered promptly in ink, in the case report forms (CRF). The principal investigator must sign the final CRF page to attest to the accuracy and completeness of the data. The data from the CRFs are then transferred to a database.

Monitoring and audit: At periods not exceeding 3 months, centers will be contacted to discuss the progress of the trial, with the purpose to verify CRF data against source records for accuracy of data recording and collection.

ELIGIBILITY:
Inclusion Criteria:

* Patient with invasive or pre-invasive (in situ) breast cancer, planned for immediate breast reconstruction post-skin sparing or nipple sparing mastectomy (unilateral or bilateral)
* Patient agrees to participate in study and to sign an informed consent form
* Able and willing to return for all scheduled and required study visits

Exclusion Criteria:

* Is a smoker (patient having quit at least 4 weeks prior surgery can be included)
* BMI <18 or > 30
* Previous radiation therapy to the region at any time
* Insulin-dependent diabetes or any immune deficiency requiring immunosuppressant use such as cortisone or biological therapies
* Predicted implant size <200 or >600 ml per investigator assessment
* Allergy to porcine
* Pregnancy or lactating
* Current enrollment or plans to enroll in another clinical trial unless a retrospective study
* Neoadjuvant treatment with chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is number of unplanned/ unanticipated surgical breast procedures. Other endpoints in the trial will be secondary. | 24 months
  Follow-up time after primary surgery is 24 months.

SECONDARY OUTCOMES:
Aesthetic outcome | 24 months
  To measure aesthetic outcome between the two study groups using a 6- point scale. The evaluation will be done by three independent groups consisting of lay people, professionals (breast/ plastic surgeons) and patient evaluation. The aesthetic evaluation will be based on the pre and postoperative photos.
Complications | 24 months
  To measure any difference between the two study groups in complication rates.
Number of surgical procedures | 24 months
  To compare the total number of surgical procedures (planned or unplanned) between the two study groups).
Cost-Benefit analysis | 24 months
  A cost-benefit analysis comparing the cost for an IBR with implant without ADM, vs. IBR with ADM (Strattice™) during a 24 months follow-up time.
Quality of Life | 24 months
  Measure Quality of Life in both groups, using the EORTC QLQ-C30 (Generic tool), EORTC-BR23 (Breast cancer specific tool), EORTC-BRR (Specific for breast reconstruction).

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Lohmander, MD, Principal Investigator — Karolinska Institutet
Locations (5):
- Sweden (4):
  - Falun Hospital, Department of Breast Surgery, Falun
  - Capio S:t Gorans Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Södersjukhuset AB, Stockholm
- Oxford University Hospitals, Oxford, United Kingdom

REFERENCES:
- [Derived] Lohmander F, Lagergren J, Johansson H, Roy PG, Brandberg Y, Frisell J. Effect of Immediate Implant-Based Breast Reconstruction After Mastectomy With and Without Acellular Dermal Matrix Among Women With Breast Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2021 Oct 1;4(10):e2127806. doi: 10.1001/jamanetworkopen.2021.27806. PMID 34596671
- [Derived] Lohmander F, Lagergren J, Johansson H, Roy PG, Frisell J, Brandberg Y. Quality of life and patient satisfaction after implant-based breast reconstruction with or without acellular dermal matrix: randomized clinical trial. BJS Open. 2020 Oct;4(5):811-820. doi: 10.1002/bjs5.50324. Epub 2020 Aug 6. PMID 32762012